CLINICAL TRIAL: NCT02294383
Title: Vaginal Tactile Imaging in Assessment of Pelvic Floor Conditions
Status: Completed | Type: Observational
Sponsor: Artann Laboratories (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: VTI05; R44AG034714 (NIH)
Record Dates: First submitted 2014-11-14; First posted 2014-11-19 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic Floor Biomechanics; Tissue Elasticity; Tactile Imaging
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Pre/post surgery pelvic floor assessment
- Conservative treatmen monitoring
- Pelvic floor muscle contrictions
- Imaging reproducibility

SUMMARY:
The clinical study includes investigation of the outcomes of surgery for biomechanical restoration of pelvic floor conditions, monitoring pelvic floor conditions under conservative treatment/management, identification and investigation changes of pelvic floor muscle contractions and their significance in characterization of pelvic floor conditions, assessment of tactile imaging reproducibility, including pelvic floor muscle contraction.

ELIGIBILITY:
Inclusion Criteria:

* No prior pelvic floor surgery, and
* Normal pelvic floor conditions, or
* POP Stage I affecting one or more vaginal compartment, or
* POP Stage II affecting one or more vaginal compartment, or
* POP Stage III affecting one or more vaginal compartment, or
* POP Stage IV affecting one or more vaginal compartment.

Exclusion Criteria:

* Active skin infection or ulceration within the vagina
* Presence of a vaginal septum;
* Active cancer of the colon, rectum wall, cervix, vaginal, uterus or bladder;
* Ongoing radiation therapy for pelvic cancer;
* Impacted stool;
* Significant pre-existing pelvic pain including levator ani syndrome, severe vaginismus or vulvadynia;
* Severe hemorrhoids;
* Significant circulatory or cardiac conditions that could cause excessive risk from the examination as determined by attending physician;
* Current pregnancy.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population comprises of patients referred to a gynecologist/urogynecologist for either regular examination or with a pelvic floor organ concern.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2014-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Tissue elasticity measured as a gradient in tactile image. Unit of Measure: kPa/mm | From 1 day to 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Princeton Urogynecology, Princeton, New Jersey
  - Institute of Female Pelvic Medicine and Reconstructive Surgery, Allentown, Pennsylvania

REFERENCES:
- [Background] Egorov V, van Raalte H, Sarvazyan AP. Vaginal tactile imaging. IEEE Trans Biomed Eng. 2010 Jul;57(7):1736-44. doi: 10.1109/TBME.2010.2045757. Epub 2010 May 17. PMID 20483695
- [Background] Egorov V, van Raalte H, Lucente V. Quantifying vaginal tissue elasticity under normal and prolapse conditions by tactile imaging. Int Urogynecol J. 2012 Apr;23(4):459-66. doi: 10.1007/s00192-011-1592-z. Epub 2011 Nov 10. PMID 22072417
- [Background] van Raalte H, Egorov V. Characterizing female pelvic floor conditions by tactile imaging. Int Urogynecol J. 2015 Apr;26(4):607-9. doi: 10.1007/s00192-014-2549-9. Epub 2014 Oct 25. PMID 25344223